CLINICAL TRIAL: NCT05993507
Title: A Scalable Psychological Intervention to Improve Mental Health Outcomes of Earthquake Survivors in Türkiye: An Open Trial Pilot Study
Brief Title: Mental Health Outcomes of Earthquake Survivors in Türkiye
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Koç University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023.214.IRB3.097
Record Dates: First submitted 2023-07-07; First posted 2023-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Mental Health Issue

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Problem Management Plus (PM+) (Experimental): As an open trial single group pre-post design, all participants in the study will receive PM+.
  Interventions: Behavioral: Problem Management Plus (PM+)

INTERVENTIONS:
Behavioral: Problem Management Plus (PM+) — Problem Management Plus (PM+) is a brief, scalable intervention that is developed by World Health Organization for communities exposed to adversity. PM+ consists of five weekly in-person sessions of 90 minutes. The intervention integrates four evidence-based behavioural strategies: arousal reduction using a slow breathing exercise (session 1), problem-solving (session 2), behavioural activation by re-engaging with pleasant and task-oriented activities (session 3) and accessing social support (session 4). Homework practice is scheduled following each session and discussed in the next session. Psychoeducation is delivered in session 1 and relapse prevention is discussed in session 5. Facilitators will receive weekly supervisions by PM+ supervisors.

SUMMARY:
The primary aim of this open trial pilot study will be to test feasibility, acceptability, and potential impact of Problem Management Plus (PM+), brief, scalable psychological intervention developed by WHO, for earthquake survivors in Türkiye. Secondly, this study aims to assess trial procedures in preparation for a future studies evaluating the effectiveness of PM+ intervention with earthquake survivors.

DETAILED DESCRIPTION:
Considering the fact that around 16% of Turkey's population is affected by the February 6 earthquakes, reaching a higher number of people on time can be achieved through the implementation of brief, scalable interventions addressing common mental health problems. This will be the first study that investigate the individual PM+ among earthquake survivors in Türkiye. Testing these interventions will provide evidence for further use in future disasters.

The study will assess changes in depression, anxiety, posttraumatic stress symptoms, psychological distress, and psychosocial functioning scores before and after the intervention. The hypothesis to be examined posits that participants will have significantly lower depression, anxiety, posttraumatic stress, psychological distress and psychosocial functioning scores at the post assessment compared to pre-assessment.

This study will be designed as a single group pre-and post-test research. The sample will be adult earthquake survivors in Türkiye. A partnership has been formed with Travma ve Afet Ruh Sağlığı Çalışmaları Derneği (TARDE), a non-governmental organization working in the earthquake-stricken regions. 30 psychologists of TARDE have been trained for PM+ for their work with people who experienced the earthquake. The outcome measures will be assessed two times: once before and once after PM+ will be conducted. After the baseline assessment, all participants will receive the consecutive 5-session on individual PM+. The PM+ intervention consists of five weekly sessions incorporating evidence-based behavioral strategies.

ELIGIBILITY:
Inclusion Criteria:

* being 18 years or above
* being experienced the earthquake
* reported elevated level of psychological distress indicated by a score of >15 on Kessler Psychological Distress Scale
* reported impaired daily functioning indicated by a score of >16 on World Health Organization Disability Assessment Scale

Exclusion Criteria:

* imminent suicide risk (assessed with the PM+ manual suicidal thoughts interview)
* severe mental disorders (e.g., psychotic disorders) or cognitive impairment (e.g., severe intellectual disability (assessed by the PM+ manual observation checklist)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-11-17 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Change of the Patient Health Questionnaire-9 (PHQ-9) over time | once before (within a few days and no longer than one week after the pre-intervention) and one week after the last session of PM+ will be conducted; which is expected to last an average of 7 weeks
  PHQ-9 is a 9 item questionnaire that measures the severity of depression symptoms. Items are scored as "0" (not at all) to "3" (nearly every day), providing a 0-27 severity score. Higher scores indicate more severe depressive symptoms.

SECONDARY OUTCOMES:
Change of the Generalized Anxiety Disorder-7 (GAD-7) over time | once before (within a few days and no longer than one week after the pre-intervention) and one week after the last session of PM+ will be conducted; which is expected to last an average of 7 weeks
  GAD-7 is a 7-item measure of general anxiety symptoms that measures anxiety symptoms. Each item is scored from 0 (not at all) to 3 (nearly every day) providing a range between 0 and 21. Higher scores indicate higher levels of anxiety.
Change of the Posttraumatic Stress Disorder Checklist for Diagnostic and Statistical Manual-5 (DSM-5) (PCL-5) over time | once before (within a few days and no longer than one week after the pre-intervention) and one week after the last session of PM+ will be conducted; which is expected to last an average of 7 weeks
  The PCL-5 is a 20-item questionnaire that assesses the symptoms of PTSD. Items are scored from 0 (not at all) to 4 (extremely) providing a range between 0 and 16. Higher scores indicate higher levels of PTSD symptoms.
Change of the Kessler Psychological Distress Scale (K-10) over time | once before (within a few days and no longer than one week after the pre-intervention) and one week after the last session of PM+ will be conducted; which is expected to last an average of 7 weeks
  K-10 is a 10-item scale that assesses the psychological distress. Each item is scored from 1 (none of the time) to 5 (all of the time) and ranges between 10 and 50. Higher scores indicate more severe psychological distress.
Change of the World Health OrganizationDisability Assessment Schedule (WHODAS 2.0) over time | once before (within a few days and no longer than one week after the pre-intervention) and one week after the last session of PM+ will be conducted; which is expected to last an average of 7 weeks
  WHODAS is a 12-item scale that assesses ability to engage in daily activities. Each item is scored from 0 (none) to 4 (extreme) and ranges between 0 and 48. Higher scores indicate more daily dysfunctioning.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşenur Coşkun Toker, MA, Study Chair — Koç University
Locations (1):
- Koc University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sangraula M, Turner EL, Luitel NP, van 't Hof E, Shrestha P, Ghimire R, Bryant R, Marahatta K, van Ommeren M, Kohrt BA, Jordans MJD. Feasibility of Group Problem Management Plus (PM+) to improve mental health and functioning of adults in earthquake-affected communities in Nepal. Epidemiol Psychiatr Sci. 2020 May 26;29:e130. doi: 10.1017/S2045796020000414. PMID 32452336
- [Background] Dawson KS, Bryant RA, Harper M, Kuowei Tay A, Rahman A, Schafer A, van Ommeren M. Problem Management Plus (PM+): a WHO transdiagnostic psychological intervention for common mental health problems. World Psychiatry. 2015 Oct;14(3):354-7. doi: 10.1002/wps.20255. No abstract available. PMID 26407793